CLINICAL TRIAL: NCT04470856
Title: Can Carotid Artery Doppler Variations Induced by End-expiratory Occlusion Manoeuvre Predict Fluid Responsiveness in Septic Shock Patients?
Brief Title: Carotid Doppler and EEOT for Fluid Responsiveness Prediction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, D'ARRIGO SONIA, principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 1677
Record Dates: First submitted 2020-07-06; First posted 2020-07-14 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Septic Shock
Keywords: end-expiratory occlusion test; septic shock; carotid doppler
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: Participants receive an 20sec-EEOT at the initial phase of the study, then they receive a fluid challenge during the second phase of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- septic shock patients (Experimental): Intubated patients with septic shock receive an end-expiratory occlusion test (EEOT) and, after the test, they receive a 500 ml-fluid challenge.
  During these phases the carotid doppler changes will be recorded.
  Interventions: Diagnostic Test: End-expiratory occlusion test (EEOT)

INTERVENTIONS:
Diagnostic Test: End-expiratory occlusion test (EEOT) — An occlusion manoeuvre during the end of expiration for 20 seconds

SUMMARY:
Fluid responsiveness prediction prior to fluid challenge administration is a topic of interest, which has been extensively investigated, but remains challenging.

In clinical practice, functional hemodynamic tests (FHT) consisting of maneuvers that affect cardiac function and/or heart-lung interaction, have been introduced in order to identify fluid responders and non-responders without fluid challenge administration.

Changes in cardiac output induced by the Passive Leg Raising (PLR) test reliably predicted the increase in cardiac output to volume expansion. New approaches have been recently developed based on changes in respiratory dynamics, such as a transient increase in tidal volume, or a lung recruitment maneuver or an end-expiratory occlusion (EEO) test. The EEO leaded to an increase in venous return, cardiac preload and stroke volume in preload-responsive patients. The authors found that an increase in cardiac output ≥ 5% during a 15-s EEO reliably predicted its response to a 500-ml saline infusion.

However, in order to identify the rapid and transient increase in cardiac index during the EEO, continuous and instantaneous cardiac output monitoring is necessary. Pulse contour analysis methods provide a beat-to-beat estimation of cardiac output and had been used in most of studies validating the EEO test.

Carotid doppler is a non-invasive, bedside, easy to use ultrasound technique that measuring blood flow peak velocity (CDPV) and duration of systolic component of each cardiac cycle (from the onset to dicrotic notch- Flow time - FT) allows a reliable estimation of fluid status and could be an interesting alternative to track changes in SV and cardiac output.

DETAILED DESCRIPTION:
The aim of the present study is to investigate whether changes in systolic peak velocity (ΔV peak-CA) and in flow time (ΔFT) using carotid artery Doppler during an End-Expiratory Occlusion Test (EEOT) predict fluid responsiveness in patients with septic shock and lung protective mechanical ventilation in ICU.

All patients will be in supine position (trunk elevated 30°), sedated, paralyzed and mechanically ventilated in the volume control mode. Tidal volume will be set at 6-8 ml/kg of predicted body weight.

They will be all monitored by an EV1000TM/Volume View (Edwards Lifesciences Corporation, Irvine, CA 92614) for measurement of cardiac index through transpulmonary thermodilution (TPTD) and pulse contour analysis. Cardiac index and the other hemodynamic parameters derived from pulse contour analysis will be continuously recorded over a 20-sec period.

Phase 1 (baseline): a first set of TPTD will be performed to assess the cardiac index (CI), the stroke volume index (SVI), the stroke volume variation (SVV), the systemic vascular resistance index (SVRI). The mean arterial pressure (MAP), heart rate (HR), central venous pressure (CVP) were also recorded. A carotid doppler was performed to measure the systolic peak velocity (CDPV) and the flow time (FT) (see below).

Phase 2 (EEOT): A 20-second EEO will be than applied through a touch of ventilator for measuring the total end-expiratory pressure. MAP, HR, SVI, CVP, SVRI, pulse contour-derived CI were averaged during the 5 last seconds of the EEO because the maximal hemodynamic effects of the occlusion were observed at this time and because the EV1000TM monitor updates the data every 20 seconds. During this pause a carotid Doppler will be performed and the last 5 seconds will be recorded.

The effects of EEOT on cardiac index will be measured by pulse contour analysis and not by TPTD because these effects must be assessed by a real-time monitoring technique. In practice, the investigators will observe the continuously changing values of pulse contour analysis-derived cardiac index while performing the Doppler measurements.

Phase 3 (fluid challenge): The patients then will receive a 10-minute infusion of 500 mL saline or lactate ringer (7 ml/kg). A last set of hemodynamic measurements, including CI, MAP, HR, SVI, CVP, SVRI, and carotid Doppler, will be recorded after fluid infusion.

As soon as the cardiac index value started to increase, the investigators will consider that it had reached its maximum. At this precise time, they will freeze the image of the echograph and performed the Doppler measurements on the values displayed during the previous seconds. If pulse contour analysis-derived cardiac index will increase ≥ 5% during the EEOT, compared to the baseline value, the patient will be consider as responder to the test.

Catecholamine's infusion, mechanical ventilation settings and bed position will be kept constant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* sedated and mechanically ventilated patients
* need a fluid challenge
* hypotension defined as a systolic arterial pressure ≤90 mmHg
* tachycardia ≥100 beats/min
* urinary flow ≤0.5 mL/kg/min for 2 hrs

Exclusion criteria:

* age< 18 y old
* significant valvular heart diseases
* cardiac arrhythmia
* peripheral arterial disease
* common carotid artery stenosis greater than 50%
* spontaneous breathing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Fluid responsiveness | during EEOT
  Evaluation of changes in systolic peak velocity (ΔV peak-CA) and in flow time (ΔFT) using carotid artery Doppler during an end-expiratory occlusion test and after fluid-challenge (500 ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinsky MR. Functional hemodynamic monitoring. Crit Care Clin. 2015 Jan;31(1):89-111. doi: 10.1016/j.ccc.2014.08.005. PMID 25435480
- [Background] Monnet X, Osman D, Ridel C, Lamia B, Richard C, Teboul JL. Predicting volume responsiveness by using the end-expiratory occlusion in mechanically ventilated intensive care unit patients. Crit Care Med. 2009 Mar;37(3):951-6. doi: 10.1097/CCM.0b013e3181968fe1. PMID 19237902
- [Background] Myatra SN, Prabu NR, Divatia JV, Monnet X, Kulkarni AP, Teboul JL. The Changes in Pulse Pressure Variation or Stroke Volume Variation After a "Tidal Volume Challenge" Reliably Predict Fluid Responsiveness During Low Tidal Volume Ventilation. Crit Care Med. 2017 Mar;45(3):415-421. doi: 10.1097/CCM.0000000000002183. PMID 27922879
- [Background] Blehar DJ, Glazier S, Gaspari RJ. Correlation of corrected flow time in the carotid artery with changes in intravascular volume status. J Crit Care. 2014 Aug;29(4):486-8. doi: 10.1016/j.jcrc.2014.03.025. Epub 2014 Apr 2. PMID 24930363
- [Background] Mackenzie DC, Khan NA, Blehar D, Glazier S, Chang Y, Stowell CP, Noble VE, Liteplo AS. Carotid Flow Time Changes With Volume Status in Acute Blood Loss. Ann Emerg Med. 2015 Sep;66(3):277-282.e1. doi: 10.1016/j.annemergmed.2015.04.014. Epub 2015 May 21. PMID 26003002
- [Background] Hossein-Nejad H, Mohammadinejad P, Lessan-Pezeshki M, Davarani SS, Banaie M. Carotid artery corrected flow time measurement via bedside ultrasonography in monitoring volume status. J Crit Care. 2015 Dec;30(6):1199-203. doi: 10.1016/j.jcrc.2015.08.014. Epub 2015 Aug 22. PMID 26410681
- [Background] Shokoohi H, Berry GW, Shahkolahi M, King J, King J, Salimian M, Poshtmashad A, Pourmand A. The diagnostic utility of sonographic carotid flow time in determining volume responsiveness. J Crit Care. 2017 Apr;38:231-235. doi: 10.1016/j.jcrc.2016.10.025. Epub 2016 Nov 9. PMID 27987483
- [Background] Ibarra-Estrada MA, Lopez-Pulgarin JA, Mijangos-Mendez JC, Diaz-Gomez JL, Aguirre-Avalos G. Respiratory variation in carotid peak systolic velocity predicts volume responsiveness in mechanically ventilated patients with septic shock: a prospective cohort study. Crit Ultrasound J. 2015 Dec;7(1):29. doi: 10.1186/s13089-015-0029-1. Epub 2015 Jun 26. PMID 26123610
- [Result] Cecconi M, De Backer D, Antonelli M, Beale R, Bakker J, Hofer C, Jaeschke R, Mebazaa A, Pinsky MR, Teboul JL, Vincent JL, Rhodes A. Consensus on circulatory shock and hemodynamic monitoring. Task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Dec;40(12):1795-815. doi: 10.1007/s00134-014-3525-z. Epub 2014 Nov 13. PMID 25392034
- [Derived] D'Arrigo S, Dell'Anna AM, Sandroni C, Messina A, Cacciola S, Pacini C, Antonelli M. Can carotid artery Doppler variations induced by the end-expiratory occlusion maneuver predict fluid responsiveness in septic shock patients? Crit Care. 2023 Apr 19;27(1):153. doi: 10.1186/s13054-023-04422-9. PMID 37076861